CLINICAL TRIAL: NCT05097742
Title: Interest of Speech Therapy in Children With Epilepsy: What Impairments of Cognitive Functions?
Brief Title: Cognitive Impairments in Children With Epilepsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0638
Record Dates: First submitted 2021-10-27; First posted 2021-10-28 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy Syndrome
Keywords: Speech therapy; Neurology; Children; Oral language; Attention; Type of epilepsy (focal epilepsy or generalized epilepsy); Etiology of epilepsy (unknown, idiopathic, structural, metabolic, immune, infectious); Epilepsy syndrome
MeSH Terms: conditions — Epileptic Syndromes; Communication Disorders; Epilepsies, Partial; Epilepsy, Generalized; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the proportion of language and attentional difficulties in patients with epilepsy is recognized, both in the literature and in the clinical experience of practitioners, it is appropriate to propose a complete speech-language assessment of oral language and attention.This study investigates these impairments through the taking of specific tests.

The general objective of this study is to observe possible oral language and attention disorders in children with epilepsy, by age and etiology of epilepsy.

The objective of this work is to study therapeutic apheresis (including plasma exchange and immunoadsorption) among french neuropediatric tertiary centers and to prove that this treatment modality is effective and well tolerated in pediatric neurology diseases.

ELIGIBILITY:
Inclusion criteria:

The subjects should :

* Be at least 3 years old and at most 15 years old
* Be French speaker
* Be in a regular class
* Have a diagnosis of epilepsy

Exclusion criteria:

* Subjects schooled in IEM
* Subjects diagnosed with austim spectrum disorder
* Subjects with a motor or visual handicap
* Subjects with psychiatric disorders

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with epilepsy followed by Dr COLMARD at the Montpellier hospital and university center
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Score in the different tests assessing oral language | day 1
  Test assessing oral language :
  * Oral naming of images
  * Oral designation of images
  * Morphosyntactic comprehension test
  * Syntactic production test
  The scores obtained in the various tests are organized into 7 classes:
  Class 1 = percentiles less than 7 : "pathological" zone Class 2 = 7 to 20 percentiles : "fragile" zone / "weak" zone Class 3 = 21 to 38 percentiles : "low standard" zone Class 4 = percentiles 39 to 62 : "median standard" zone / expected average results for age or grade level Class 5 = 63 to 80 percentiles : "higher standard" zone Classes 6 and 7 = respectively 81 to 93 percentiles and percentiles greater than 93 : zone with results well above the norm for age or grade level.

SECONDARY OUTCOMES:
Score in the different tests assessing attention | day 1
  Tests assessing attention :
  * Visual attention test
  * Auditive attention test
  The scores obtained in the various tests are organized into 7 classes:
  Class 1 = percentiles less than 7 : "pathological" zone Class 2 = 7 to 20 percentiles : "fragile" zone / "weak" zone Class 3 = 21 to 38 percentiles : "low standard" zone Class 4 = percentiles 39 to 62 : "median standard" zone / expected average results for age or grade level Class 5 = 63 to 80 percentiles : "higher standard" zone Classes 6 and 7 = respectively 81 to 93 percentiles and percentiles greater than 93 : zone with results well above the norm for age or grade level.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime colmard, résident, Principal Investigator — UH MONTPELLIER; Moritz-Gasser Sylvie, Study Chair — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC